CLINICAL TRIAL: NCT01318759
Title: (MIGA) Mini Geriatric Assessment as Compared to the Current CGA
Brief Title: (MIGA) Mini Geriatric Assessment To Replace the Comprehensive Geriatric Assessment
Acronym: MIGA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Yaffa Lerman MD, Tel-Aviv Sourasky Medical Center
Other Study IDs: 0047-11-tav
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-03

CONDITIONS: Geriatric Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a comprehensive Geriatric Assessment (CGA) currently used to evaluate elderly people in order to be able to assess their multiple organ pathology, cognitive, functional and social problems. This CGA is a very time consuming tool although a powerful one.

The investigators want to present a new assessment test witch is short and comprehensive tool witch will be checked in ambulatory and in-hospital geriatric patients.

DETAILED DESCRIPTION:
MIGA test (Mini Geriatric Assessment) includes the following parameters Walking outdoors, Transfer, ADL-Dressing, Washing, Continence, Vision, Hearing, Pain, Sleeping, Weight loss, Get-Up-And-Go test, Short term memory, Clock drawing test, Falls, functional reach of hands, Depression, Behavioral problems, social support, Admissions, Polypharmacy,

All patients will be assessed by the traditional CGA and by the new MIGA test. Time consuming of the two tests will be measured and compared.

ELIGIBILITY:
Inclusion Criteria:

* Elderly people age 65 and above,
* In patients hospitalized in the geriatric department
* Out patients -from the geriatric out patient clinic
* Elderly patients visiting in the emergency room

Exclusion criteria:

* People under 65 years old
* Critically ill patients ( acute infection, acute myocardial infarction, hypoxia, hemodynamic instability)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: people aged over 65
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yaffa Lerman, MD, Study Director — Tel-Aviv Sourasky Medical Center; Oksana Borodin, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Geriatric department , Tel Aviv Sourasky Medical Center, Tel Aviv, Israel